CLINICAL TRIAL: NCT06702670
Title: Anticholinergics for Cervical Edema in Labor (ACCEL)
Brief Title: Anticholinergics for Cervical Edema in Labor
Acronym: ACCEL
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Samantha Antonioli, Resident, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-24-0841
Record Dates: First submitted 2024-11-20; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Labor Dystocia
Keywords: dilation; labor
MeSH Terms: conditions — Dystocia; Dilatation, Pathologic | interventions — Therapeutics; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with Diphenhydramine (Experimental)
  Interventions: Drug: Treatment with Diphenhydramine; Combination Product: Usual Care
- Usual Care (Active Comparator)
  Interventions: Combination Product: Usual Care

INTERVENTIONS:
Drug: Treatment with Diphenhydramine — Diphenhydramine 50mg IV will be administered within 1 hour of the cervical exam which diagnosed prolonged active phase of labor
  Arms: Treatment with Diphenhydramine
Combination Product: Usual Care — Participants will receive cervical exams every 2 hours in active labor, placement of intrauterine pressure catheter, up titration of Pitocin if contractions are inadequate, maternal repositioning, and use of adjunct devices such as a peanut ball.

SUMMARY:
The purpose of this study is to is to determine the clinical effectiveness of a single dose of intravenous (IV) medication for the prevention of labor arrest and cesarean delivery in primiparous women undergoing trial of labor.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous
* Viable single intrauterine pregnancy

  -≥ 34 weeks of gestation
* Ruptured membranes
* Category I tracing at time of inclusion
* Active phase of labor (>=6 cm of cervix dilation)

Exclusion Criteria:

* Category II or III tracing
* Allergy to the study medication (IV Diphenhydramine)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants that achieve complete dilation of cervix (10cm) | from start of treatment upto 4 hours
Number of participants that achieve complete dilation of cervix (10cm) | from start of treatment upto 6 hours

SECONDARY OUTCOMES:
Number of participants who have vaginal delivery after protracted labor | End of delivery (an average of upto 6 hours after start of treatment)
Number of participants who have Postpartum complications captured as composite maternal morbidity | from hospitalization up to 6 weeks postpartum
  This includes postpartum hemorrhage, cervical lacerations or intraamniotic infection
Number of neonates that had adverse events | from birth up to 6 weeks post-delivery
  Adverse events include 5 minute APGAR SCORES less than 7, Respiratory Support with intubation in the delivery room , Neonatal intensive acre unit (NICU) admission, Fetal Anomalies, Infection, Intraventricular Hemorrhage, Hypoglycemia, Retinopathy of prematurity, Injuries, Fractures

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Antonioli, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No